CLINICAL TRIAL: NCT05341310
Title: A Virtual Clinic for Parents of Children With ADHD - an Individually-tailored Approach to Reduce Parental Distress
Brief Title: An Internet-delivered Intervention for Parents of Children With ADHD
Acronym: ADHDCoach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Costina-Ruxandra Poetar, Assistant professor, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PN-III-P1-1.1-PD-2019-1191
Record Dates: First submitted 2022-04-11; First posted 2022-04-22 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: ADHD
Keywords: Internet intervention; individually-tailored intervention; parental distress; ADHD; children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADHDCoach (Experimental): Participants in the experimental group will have access to an individually-tailored Internet intervention developed for the present study. The intervention in clinician-guided and it consists of nine modules delivered for four weeks. The Internet Intervention, called ADHDCoach, is based on an existent Behavioral Parent training protocol, an intervention that was previously tested in a randomized controlled trial with Romanian children. The contents for parent modules were developed according to Rational Emotive and Behavioral Therapy.
  Interventions: Behavioral: ADHDCoach; Other: Treatment as usual
- Treatment as usual (Active Comparator): Treatment as usual at the outpatient clinic
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: ADHDCoach — ADHDCoach is an individually-tailored intervention to reduce parents' of children diagnosed with ADHD distress.
  Arms: ADHDCoach
Other: Treatment as usual — Treatment as usual in the outpatient clinic

SUMMARY:
The aims of the present study is to investigate the efficacy of a co-designed individually-tailored Internet intervention for parents of children with ADHD.

DETAILED DESCRIPTION:
Attention/deficit-hyperactivity disorder is a prevalent mental health problem in children with a significant impact on children, families and society. Despite the fact that evidence-based treatment exists, with pharmacologic and non-pharmacologic options available, a significant percentage of children do not have access to treatment. Behavioral parent training is recommended as first line treatment for children with ADHD, however, parents face numerous challenges in access, and even when they access BPT, dropout rates are high. Technology could improve access to evidence-based treatments and surpass existent gaps. For instance, Internet interventions are associated with moderate to large effect sizes for anxiety and depressive symptoms in adults.

Participants included in this study, namely parents of children diagnosed with ADHD (aged 6-11 years) will be randomized either to ADHDCoach intervention or Treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child diagnosed with ADHD
* Child aged between 5-11 years
* Have Internet access
* Have ability to read and write in Romanian
* No medication/ or stable dose of pharmacological treatment

Exclusion Criteria:

* Other ongoing psychological treatment or counselling for mental health problems (currently undergoing psychotherapy or participating in a parenting program for child ADHD)
* Recent (within the past 3 months) changes in the dose of medication
* Serious psychopathology requiring immediate clinical attention (e.g., severe depressive symptoms)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Changes in parental psychological distress | Baseline, 4 weeks and follow-up at 3 months after treatment termination
  The Patient Health Questionnaire will be used to assess changes in parental anxiety and depressive symptoms from pre-treatment to post-treatment and follow-up. Scores range between 0 and 12, higher scores indicate higher anxiety and depressive symptoms.

SECONDARY OUTCOMES:
Changes in child ADHD symptoms | Baseline, 4 weeks and follow-up at 3 months after treatment termination
  The ADHD Rating Scale-5 Home version is a 18 items scale measuring Inattention and Hyperactivity in children. Scores range from 0 to 54, higher scores indicate higher ADHD symptoms.
Changes in parenting | Baseline, 4 weeks and follow-up at 3 months after treatment termination
  The Alabama Parenting Questionnaire- short form consists of 9 items rated on a 5 points Likert scale (1 - Never, 5 - Always). Scores will be reported for positive parenting, poor monitoring and inconsistent discipline. For each subscale, scores range between 1 and 15. Higher scores for positive parenting subscale indicate higher positive parenting practices, while higher scores for poor monitoring and inconsistent discipline indicate higher negative parenting practices.
Changes in parent-child closeness | Baseline, 4 weeks and follow-up at 3 months after treatment termination
  Parent-child closeness will be measured via three items in line with previous research. Answers are rated on a 5-point Likert scale, ranging from 1 (Never) to 5 (Always). Scores range from 0 to 15, higher scores indicate higher parent-child closeness.
ADHD adult | Baseline, 4 weeks and follow-up at 3 months after treatment termination
  The Adult Self-Report Screening Scale for DSM-5 consists of 6 items, rated on a 5 points Likert scale (0 - Never, 4 - Very often). Scores range from 0 to 24. Higher scores indicate higher ADHD symptoms.
Changes in ADHD Knowledge | Baseline, 4 weeks and follow-up at 3 months after treatment termination
  A knowledge test regarding ADHD symptoms, causes and treatment was developed for the presents study. The scale consists of 15 items with a True or False choice. Scores are also rated on the certainty of the answers provided. Total scores range from 0 to 15. Higher scores indicate a better knowledge regarding ADHD.
Satisfaction with the intervention | At 4 weeks after treatment initiation
  Client Satisfaction Questionnaire-8. Scores range between 0 and 32, higher scores indicate higher satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Costina R Păsărelu, Ph.D, Principal Investigator — Babes-Bolyai University
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No